CLINICAL TRIAL: NCT03445598
Title: A Novel and Adaptive Software for Automated Delivery of Cognitive Behavioral Therapy
Brief Title: Automated and Personalized Cognitive Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indian Institute of Technology Kanpur (Other)
Responsible Party: Principal Investigator, Nitin Gupta, Assistant Professor, Indian Institute of Technology Kanpur
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IITK/NG/CBT1
Record Dates: First submitted 2018-02-14; First posted 2018-02-26 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Depressive Symptoms
Keywords: depression; anxiety; CBT; psychotherapy; e-health; CCBT
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant is masked to the intervention assigned to them. All outcome measures are self-reported by the participants through a computer program without any involvement of the experimenters.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive CCBT group (Experimental): This group receives Interactive and Personalized CCBT
  Interventions: Behavioral: Interactive and personalized CCBT
- Limited CCBT control group (Active Comparator): This group receives Feature-limited CCBT
  Interventions: Behavioral: Feature-limited CCBT
- Waitlist control group (Other): This group receives waitlist control
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: Interactive and personalized CCBT — Participants will go through an automated program. Participants will learn and practice the techniques of CBT through multimedia elements along with personalized content and interactive features in the program
  Arms: Interactive CCBT group
Behavioral: Feature-limited CCBT — Participants will be going through an automated program. Participants will learn and practice the techniques of CBT in a plain-text format with reduced features.
  Arms: Limited CCBT control group
Other: Waitlist control — Participants will be put on a waitlist for a period of 6 weeks.
  Arms: Waitlist control group

SUMMARY:
This study is designed to evaluate a novel online tool to deliver computerized Cognitive Behavioral Therapy (CBT). Participants will be randomized into three groups: experimental, active control, and waitlist. Participants in the experimental group will have access to the full-featured online tool designed to deliver CBT in an interactive and personalized manner. The participants in the active control group will have access to a limited version of the online tool designed to deliver basic CBT in plain text format. The waitlisted participants will be put on a waitlist for 6 weeks. We hypothesize that the experimental group participants will show a significantly higher reduction in depression symptom severity and will show increased engagement and adherence to the online tool.

DETAILED DESCRIPTION:
Depression is a major psychiatric disorder globally, including in India. One of the most effective approaches to treat depression is Cognitive Behavioral Therapy (CBT), but its reach is limited by the dearth of trained psychiatrists, especially in remote areas, and the high costs and stigma associated with visits to a psychiatric clinic. Delivering CBT through a computer, with limited or no intervention from a psychiatrist, could address these limitations. Computerized Cognitive Behavioral Therapy (CCBT) is thus emerging as a more accessible and economical alternative to CBT. Despite some evidence of its efficacy, CCBT use is limited because the existing software programs used to deliver the therapy provide a much lower level of personalization and engagement than in-person therapy. The objective of this study is to assess if the new algorithm makes CCBT more efficacious, acceptable and engaging to users. Depression severity as measured by the Patient Health Questionnaire-9 (PHQ-9) is expected to reduce over the duration of the study, more significantly in the treatment group compared to the control group. Participants will be recruited online through a website that will check compatibility with inclusion/exclusion criteria and get the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* PHQ-9 Score from 5 to 19
* Access to internet-connected computer or tablet device
* Country: India

Exclusion Criteria:

* Suicide ideation (score greater than 0 on the 9th question of PHQ-9)
* Unemployed
* Current or previous diagnosis of bipolar disorder/manic-depressive disorder or psychosis
* Prospective participants who say they only want to check out the program and do not plan to complete it are excluded.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 score | change from baseline to program completion or last usage (upto 90 days).
  Standard questionnaire for depressive symptoms. Total score is used; lower score indicates better outcome.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder 7 score | baseline, post-completion or last usage (upto 90 days), 90 day follow-up after completion
  Standard questionnaire for generalized anxiety symptoms. Total score is used; lower score indicates better outcome.
Time spent with the program | from beginning till last usage (upto 180 days)
  Automated measure of time spent on the program for experimental and active comparator group
Follow-up Patient Health Questionnaire-9 score | 90 days after program completion
  Standard questionnaire for depressive symptoms. Total score is used; lower score indicates better outcome.

OTHER OUTCOMES:
Change in Patient Health Questionnaire-9 score (Intermediate reports) | after modules 1 (average 1 week), 2 (average 2 weeks), 3 (average 3 weeks), 4 (average 4 weeks) and 5 (average 5 weeks)
  Standard questionnaire for depressive symptoms. Total score is used; lower score indicates better outcome.
Change in Generalized Anxiety Disorder 7 score (Intermediate reports) | after modules 1 (average 1 week), 2 (average 2 weeks), 3 (average 3 weeks), 4 (average 4 weeks) and 5 (average 5 weeks)
  Standard questionnaire for generalized anxiety symptoms. Total score is used; lower score indicates better outcome.
User experience survey | after module 3 (average 3 weeks) and module 6 (upto 90 days) of program
  Computerized survey to get user feedback on the features of the program
Change in Patient Health Questionnaire-9 score (for clinician-referred participants) | baseline, post-completion or last usage (upto 90 days), 90 day follow-up after completion
  The subset of participants that are referred to the trial by a clinician can be analyzed separately to test the effectiveness of the program when used with a clinician's referral. Total score is used; lower score indicates better outcome.
Change in Generalized Anxiety Disorder 7 score (for clinician-referred participants) | baseline, post-completion or last usage (upto 90 days), 90 day follow-up after completion
  The subset of participants that are referred to the trial by a clinician can be analyzed separately to test the effectiveness of the program when used with a clinician's referral. Total score is used; lower score indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Gupta, PhD, Principal Investigator — Indian Institute of Technology Kanpur
Locations (1):
- Indian Institute of Technology Kanpur, Kanpur, Uttar Pradesh, India

REFERENCES:
- [Background] Gilbody S, Brabyn S, Lovell K, Kessler D, Devlin T, Smith L, Araya R, Barkham M, Bower P, Cooper C, Knowles S, Littlewood E, Richards DA, Tallon D, White D, Worthy G; REEACT collaborative. Telephone-supported computerised cognitive-behavioural therapy: REEACT-2 large-scale pragmatic randomised controlled trial. Br J Psychiatry. 2017 May;210(5):362-367. doi: 10.1192/bjp.bp.116.192435. Epub 2017 Mar 2. PMID 28254959
- [Background] Gilbody S, Littlewood E, Hewitt C, Brierley G, Tharmanathan P, Araya R, Barkham M, Bower P, Cooper C, Gask L, Kessler D, Lester H, Lovell K, Parry G, Richards DA, Andersen P, Brabyn S, Knowles S, Shepherd C, Tallon D, White D; REEACT Team. Computerised cognitive behaviour therapy (cCBT) as treatment for depression in primary care (REEACT trial): large scale pragmatic randomised controlled trial. BMJ. 2015 Nov 11;351:h5627. doi: 10.1136/bmj.h5627. PMID 26559241
- [Derived] Ghosh A, Cherian RJ, Wagle S, Sharma P, Kannan KR, Bajpai A, Gupta N. An Unguided, Computerized Cognitive Behavioral Therapy Intervention (TreadWill) in a Lower Middle-Income Country: Pragmatic Randomized Controlled Trial. J Med Internet Res. 2023 Apr 26;25:e41005. doi: 10.2196/41005. PMID 37099376
- See also: Online recruitment page — https://www.treadwill.org/iitk